CLINICAL TRIAL: NCT06676761
Title: Outcomes of a Novel Technique Minimal Scar Mastectomy
Status: Recruiting | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRB 2020/2147
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: breast cancer; nipple sparing mastectomy
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Subcutaneous; Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- nipple sparing mastectomy without reconstruction: nipple sparing mastectomy without reconstruction
  Interventions: Procedure: nipple sparing mastectomy without reconstruction

INTERVENTIONS:
Procedure: nipple sparing mastectomy without reconstruction — nipple sparing mastectomy was conventionally performed with reconstruction. we aim to study the outcomes in the group of patients with Minimal scar mastectomy (MSM) who have nipple sparing mastectomy without reconstruction

SUMMARY:
Nipple sparing mastectomy is oncologically safe and has a good cosmetic outcome. However, nipple sparing mastectomy was conventionally performed with reconstruction. Minimal scar mastectomy (MSM) is a novel technique which could allow women, with non-ptotic breasts, who do not want reconstruction, to conserve their nipple areolar complex (NAC) and avoid the transverse scar associated with modified radical mastectomy. This is the first study on the oncologic and surgical outcomes of MSM.

ELIGIBILITY:
Inclusion Criteria: breast cancer patients who opted for minimal scar mastectomy -

Exclusion Criteria: breast cancer patients who underwent conventional mastectomy

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — female breast cancer patients
Study Population: breast cancer patients with non-ptotic breasts, who do not want reconstruction, to conserve their nipple areolar complex (NAC) and avoid the transverse scar associated with modified radical mastectomy.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
oncological outcome | 5 years from operation
  recurrence rate

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided
will consider sharing IPD when paper was accepted for publication

REFERENCES:
- [Background] Lim GH, Allen JC, Ng RP. Oncoplastic round block technique has comparable operative parameters as standard wide local excision: a matched case-control study. Gland Surg. 2017 Aug;6(4):343-349. doi: 10.21037/gs.2017.03.06. PMID 28861374
- [Background] Lim GH. How to do minimal scar mastectomy: first-reported novel concept of nipple sparing mastectomy without reconstruction. ANZ J Surg. 2018 Dec;88(12):1345-1346. doi: 10.1111/ans.14941. Epub 2018 Nov 1. No abstract available. PMID 30384398